CLINICAL TRIAL: NCT05372094
Title: Noise Reduction Preferences in Teenagers and Pre-teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-802
Record Dates: First submitted 2022-05-03; First posted 2022-05-12 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: All participants will be fit with hearing aids with the same noise reduction feature. This feature has distinct, discrete levels of noise reduction which will be evaluated by the participants.
Masking Description: Participants will be blinded as to which noise reduction setting they are listening to during lab visit objective testing only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): Participants will be fit with a commercially available hearing aid and tested using various strengths of the noise reduction feature.
  Interventions: Device: Phonak Hearing Aid

INTERVENTIONS:
Device: Phonak Hearing Aid — Commercially available hearing aid with various noise reduction strengths

SUMMARY:
Noise reduction preferences and blue tooth access to hearing aid streaming features will be evaluated in experienced hearing aid users age 10-17.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the preferences for hearing aid noise reduction settings in users age 10 -17, as well as to evaluate preferences for accessing the hearing aid Bluetooth streaming programs for this population. Subjective preferences will be obtained by having the participants listen to a noisy scene with different levels of noise reduction, to which they are blinded, and rate their preference. Blinded objective speech performance testing will be completed by a) finding the signal-to-noise ratio at which participant can correctly repeat back 50% of the target words, and b) measuring the percent of words correctly repeated during a noisy listening task. These tasks will be done using different levels of noise reduction. Subjective preferences for accessing Bluetooth streaming will also be obtained by asking participants which method they prefer (phone, hearing aid, or touch control).

.

ELIGIBILITY:
Inclusion Criteria:

* mild, moderate, or moderate-severe bilateral sensorineural hearing loss
* native English speakers with ability to communicate verbally
* able to read and follow directions
* access to smartphone and willing to download a hearing aid app
* experienced hearing aid user (6+ months)

Exclusion Criteria:

* unable to follow verbal directions
* unable to communicate verbally
* unable to wear study devices for required home trials
* active middle ear infection
* unable to attend lab visits required for study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 14.33 [10 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Listening Effort Questionnaire
Description: Participant will rate perceived listening effort during a speech in noise task with different levels of noise reduction. Participants will rate how easy the task seemed using a sliding scale with 100 increments between two verbal anchors: "it was very easy" to "it was not easy at all". Higher scores indicate higher perceived listening effort. A rating of "0" would indicate "it was very easy" to understand the speech while a rating of "100" would indicate "it was not easy at all" to understand the speech.
Time Frame: Day 14 of study, visit 2
Population: All participants who completed the testing except three identified outliers (two who never wore hearing aids and one who was not able to complete activities assigned during the home trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 15
units on a scale
  Subjective rating with NR OFF | 44.73 (27.54)
  Subjective rating with NR at custom setting | 44.5 (27.45)
  Subjective rating with NR at WEAK | 41.53 (26.7)
  Subjective rating with NR at STRONG | 35.86 (26.91)
Statistical Analysis 1: Comparison: Experimental; Fixed factor of program and random intercept of participant; Test type: Other; p = 0.007, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental; Follow up comparison between noise reduction setting OFF and noise reduction setting STRONG; Test type: Other; p < 0.05, Mixed Models Analysis
Statistical Analysis 3: Comparison: Experimental; Follow up comparison between noise reduction setting STRONG and noise reduction setting WEAK; Test type: Other; p < 0.01, Mixed Models Analysis
Statistical Analysis 4: Comparison: Experimental; Follow up comparison between ratings of effort with "OFF" and "WEAK"; Test type: Other; p > .05, Mixed Models Analysis

2. Secondary Outcome: Speech Reception Threshold
Description: The signal to noise ratio in which participant can correctly repeat 50% of key words at different levels of noise reduction, known as SNR50. A lower number is better, as it indicates that the words do not have to be presented at a much higher level than the noise in order for the person to understand 50% of the words. For example, an SNR of 2 dB means that the words are 2 dB louder than the noise, and SNR of 0 dB means that the words and the noise are at the same level, etc.
Time Frame: Day 28, visit 3
Population: All participants who completed the task except three identified outliers.
Measure: Mean (Full Range); unit: decibels (dB)
Arm/Group | Experimental
Number analyzed (Participants) | 15
decibels (dB)
  SNR50 with NR setting OFF | 1.01 [0.92 to 1.13]
  SNR50 with NR setting WEAK | 1.02 [0.95 to 1.17]
  SNR50 with NR setting MODERATE | 1.02 [0.95 to 1.14]
  SNR50 with NR setting at STRONG | 1.02 [0.94 to 1.17]
Statistical Analysis 1: Comparison: Experimental; Test type: Other; p = 0.283, Mixed Models Analysis

3. Secondary Outcome: Physical Response Time
Description: Length of time(in milliseconds) it takes participant to respond physically by pressing a button while also performing a verbal task. Participants repeat the word they hear, while at the same time, are instructed to press a button if the word they hear is an object "bigger than a basketball". A higher response time may indicate increased listening effort.
Time Frame: Day 14 of study, visit 2
Population: All participants who were able to complete the task excluding three outliers who were excluded from all analyses and one participant who was unable to perform this task.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Experimental
Number analyzed (Participants) | 14
milliseconds
  Response time with NR OFF | 2452.65 (561.43)
  Response time with NR WEAK | 2432.16 (509.75)
  Response time with NR STRONG | 2388.25 (468.62)
  Response time with NR at a custom setting | 2367.7 (448.7)
Statistical Analysis 1: Comparison: Experimental; Analysis was done only between NR OFF and NR at a custom or preferred setting; Test type: Other; p = 0.145, Mixed Models Analysis

4. Secondary Outcome: Subjective Preference Questionnaire for Hearing Aid Noise Reduction Settings
Description: A blinded paired comparison between two different settings of noise reduction (NR), while listening to a story presented in noise. Participants indicate whether they prefer listening to setting "A" or setting "B". Investigator will switch the settings so that participant is not aware of what the settings are. There will be a total of 18 trials; 12 which will compare OFF to either WEAK or STRONG, and six trials will compare WEAK to STRONG. The preferred setting will be determined by counting which setting is chosen most often from those six trials. The outcome measure data will report a count of participants who preferred OFF to their chosen setting, who preferred their chosen setting to OFF, and those who chose OFF and their preferred setting an equal number of times.
Time Frame: Day 1 of study, visit 1
Population: All participants who completed the task excluding three identified outliers who were excluded from all analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 15
Participants
  Preferred NR off | 1
  Preferred NR at individual preferred setting | 5
  Preferred OFF and preferred setting the same | 9
Statistical Analysis 1: Comparison: Experimental; An exact binomial test was performed to evaluate if the majority of teens and pre-teens with mild to severe hearing loss preferred NR setting (i.e., either weak or strong) to the NR setting OFF; Test type: Other; p = 0.3018, Exact Binomial test

5. Secondary Outcome: Subjective Questionnaire on Preference for Accessing Bluetooth on Phone
Description: Subjective questionnaire about streaming access preferences. Participants will indicate which method (Hearing aid push button, phone control, or tap control on hearing aid) for answering phone calls and listening to audio streaming on phone.
Time Frame: Day 28, visit 3
Population: All participants who completed testing excluding three identified outliers and one participant who did not use Tap Control during the home trial period.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 14
Participants
  Prefer tapping to access streaming over using phone controls or hearing aid button | 10
  Prefer tapping to answer phone call over using phone or hearing aid button | 8
  Prefer tapping to access voice assistant over using phone control or hearing aid button | 6
Statistical Analysis 1: Comparison: Experimental; Exact binomial test was done to evaluate if the majority (>50%) of teens and pre-teens prefer to use Tap Control to access Bluetooth streaming, compared to using the HA push button or phone controls; Test type: Other; p = 0.1796, Exact Binomial test

6. Secondary Outcome: Verbal Response Accuracy
Description: Out of 25 monosyllabic words presented in noise at different levels of noise reduction, the number of words the participant correctly repeats,while also performing a visual task. No statistical analysis was performed for this test.
Time Frame: Day 14 of study, visit 2
Population: All participants who completed the task excluding three identified outliers who were excluded from all analyses.
Measure: Mean (Full Range); unit: words repeated correctly
Arm/Group | Experimental
Number analyzed (Participants) | 15
words repeated correctly
  Noise Reduction setting OFF | 14.37 [7.5 to 18]
  Noise Reduction setting WEAK | 14.17 [8 to 19]
  Noise Reduction setting STRONG | 13.93 [6 to 18]
  NR setting CUSTOM | 14.3 [7.5 to 18]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT05372094/Prot_SAP_000.pdf